CLINICAL TRIAL: NCT06138314
Title: A Feasibility and Acceptability Study of a Physical Exercise Program Including Neural Mobilization to Improve Pain, Functional Status, and Physical Performance in Older Adults With Chronic Musculoskeletal Pain
Brief Title: A Pilot Study of a Neural Mobilization Intervention Applied to Older Adults With Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Frederico Mesquita Baptista, Principal Investigator, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT1
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Chronic Musculoskeletal Pain; Chronic Pain; Chronic Musculoskeletal Disease; Older Adults
Keywords: elderly; physical therapy; neural mobilization
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group will perform a physical exercise program twice a week for a period of 8 weeks.
  Interventions: Other: Physical Exercise Program
- Experimental group (Experimental): The experimental group will perform the same physical exercise program performed by participants in the control group, in addition to neural mobilization techniques twice a week for a period of 8 weeks.
  Interventions: Other: Physical Exercise Program; Other: Neural Mobilization

INTERVENTIONS:
Other: Physical Exercise Program — The physical exercise program will consist of exercises from three different exercise modalities: aerobic training, balance exercises, and isometric exercises.
Other: Neural Mobilization — Neural mobilization techniques for the upper and lower quadrants will be actively performed by participants.
  Other Names: Neurodynamics
  Arms: Experimental group

SUMMARY:
The goal of this pilot study is to evaluate the feasibility of integrating neural mobilization techniques into a multimodal physical exercise program for older adults with chronic musculoskeletal pain. The main questions it aims to answer are:

* What is the average time to assess secondary outcomes for each participant?
* What proportion of participants adhered and/or withdrew from the study at the end of the intervention protocol?
* Are there adverse events/effects associated with the intervention protocol?
* What is the level of approval/satisfaction of the participants in relation to the assessment and intervention protocols?
* What is the impact of the intervention protocol on participants´ pain, function, physical performance, somatosensory function, and nerve excursion (secondary outcomes)?

Participants will be assessed at 3 different moments: initial assessment (T0), at the end of the intervention protocol (8 weeks) (T1) and 3 months after the end of the intervention protocol (T2). The intervention protocol will consist of a multimodal exercise program (with or without integration of neural mobilization techniques) to be carried out over a period of 8 weeks at a frequency of twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 60 years or older, with primary or secondary chronic musculoskeletal pain in any body site and able to walk independently

Exclusion Criteria:

* Individuals with post-surgical pain as a result of surgery performed in the last 6 months;
* Patients with a self-reported diagnoses of infection diseases, dementia, tumor/cancer, neurodegenerative diseases, stroke, uncontrolled diabetes, or at high risk of developing cardiovascular events;
* Those with physical limitations that make it impossible for them to carry out the intervention protocols independently (e.g., wheelchair user);
* Patients who are receiving another physical therapy intervention to treat their pain.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
Dropout and adherence rates | T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Proportion of participants who adhered and withdrew from the study at the end of the intervention protocol. "Adherence to treatment" will be considered if the participant attends at least 12 sessions (75% of the total scheduled sessions).
Adverse events and adverse effects | T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Proportion of participants that reported adverse events and adverse effects during the intervention protocol.
Practicality | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  The average time taken to assess secondary outcomes for each participant.
Acceptability | T1: 8 weeks (post-intervention assessment)
  The degree to which participants approve of or are satisfied with the assessment and intervention protocols. Acceptability will be assessed qualitatively through focus groups, where a recorded interview (audio only) will be carried out by the study's main researcher, in order to assess the participants' perception of the study and the intervention protocol.

SECONDARY OUTCOMES:
Pain severity | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Brief Pain Inventory (BPI)
Temporal characteristics of pain | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  World Health Organization (WHO) Classification - It is a categorical variable with three different possible response categories:
  * Episodic recurrent pain - recurrent pain attacks with pain-free intervals;
  * Continuous pain - pain is always present;
  * Continuous with pain attacks - recurrent pain flare-ups as exacerbations of ongoing underlying pain.
Neuropathic pain components | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  painDETECT questionnaire - The instrument consists of 4 sections related to: (1) pain intensity in the last 4 weeks; (2) the pain pattern; (3) regions of pain; and (4) presence of neuropathic descriptors. The total score is obtained by adding the scores of the last 3 sections and can vary from 1 to 38. Scores ≤ 12 = the neuropathic mechanism is very unlikely to be present (predominance of the nociceptive mechanism); Scores ≥ 19 = there is a high probability of a predominant neuropathic mechanism; Scores > 12 and < 19 = the presence of a mixed component.
Pain Catastrophizing | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Pain Catastrophizing Scale (PCS) - The instrument has 13 items subdivided into three different subscales: helplessness (items 1, 2, 3, 4, 5, and 12); magnification (items 6, 7, and 13); and rumination (items 8, 9, 10, and 11). All subscales are evaluated on a 5-point Likert scale, from 0 (not at all) to 4 (all the time), where higher scores represent a greater level of catastrophizing.
Fear of Movement | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Tampa Scale for Kinesiophobia - The instrument comprises 13 items rated on a 4-point Likert scale, as follows: (1) strongly disagree; (2) somewhat disagree; (3) somewhat agree; (4) strongly agree. The higher the score, the greater the fear perceived during the execution of the movement.
Symptoms of Central Sensitization | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Central Sensitization Inventory (CSI)
Pressure Pain Threshold (Thenar region of the right hand; Right calcaneus; Region of greatest pain) | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Algometer
Cold and Warm Perception Threshold ((Thenar region of the right hand; Right calcaneus; Region of greatest pain) | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Q-sense
Lower Limb Strength | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Five Times Sit to Stand Test
Grip Strength | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Hand-held dynamometer
Agility and Dynamic Balance | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Timed-Up-And-Go Test
Nerve excursion (median and tibial nerves) | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Ultrasonography - The longitudinal and transverse excursion of the tibial and median nerves will be measured in millimeters using ultrasound images taken during the execution of a joint movement.
Range of Motion (ankle dorsiflexion and wrist extension) | T0: baseline assessment; T1: 8 weeks (post-intervention assessment); T2: 3 months post-intervention (follow-up assessment)
  Goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aveiro, Aveiro, Portugal